CLINICAL TRIAL: NCT00158808
Title: Assess the Immunogenicity &d Reactogenicity of a Booster Dose of a Formulation of GSK Biologicals' DTPw-HBV/Hib Vaccine at 15-18 Mths of Age in Infants Previously Primed With the Same Vaccine
Brief Title: Immune Memory Foll Pry Vaccination With DTPw-HBV/Hib Vaccine Formulation; Immuno & Reacto of Booster Dose at 15-18 Mths
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 101477
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hib Disease; Hepatitis B; Pertussis; Prophylaxis of Diphtheria; Tetanus
MeSH Terms: conditions — Hepatitis B; Whooping Cough; Tetanus | interventions — Tetanus Toxoid; Hepatitis B Vaccines

INTERVENTIONS:
Biological: Diphteria, tetanus, whole-cell pertussis, hepatitis B & Hib

SUMMARY:
To assess the anti-PRP antibody response one month after vaccination in the groups receiving a fourth consecutive dose of two formulations of DTPw-HBV/Hib vaccine

DETAILED DESCRIPTION:
All subjects were previously primed with one of the two formulations of the combined DTPw-HBV/Hib vaccine. At the age of 10 months, 50% of each group received a plain PRP challenge to assess the immune memory to PRP. In this booster study in the second year of life, all subjects who received DTPw-HBV/Hib and plain PRP will receive DTPw-HBV as a booster vaccination. All other subjects will receive as booster the same vaccine they received in the primary vaccination study.

ELIGIBILITY:
Inclusion criteria

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female of at least 15 months of age at the time of the booster vaccination, who had previously received 3-dose primary vaccination and, if applicable, plain-PRP vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering the study.

Exclusion criteria for enrolment

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before and ending 30 days after administration of study vaccines with the exception of oral polio vaccine (OPV).
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster dose.
* Previous booster vaccination against diphtheria, tetanus, pertussis, hepatitis B or Hib with the exception of plain PRP challenge.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.

Min Age: 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2005-01; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Anti-PRP antibody concentration one month after the booster dose (in groups boosted with the DTPw-HBV/Hib vaccine).

SECONDARY OUTCOMES:
Immunology
At the time of the booster dose: concentrations of antibodies against all vaccine antigens (diphtheria, tetanus, pertussis, hepatitis B and Hib antigens)
One month after the booster dose: concentrations of antibodies against all vaccine antigens (diphtheria, tetanus, pertussis, hepatitis B and Hib antigens)
Reactogenicity and Safety
Occurrence of solicited symptoms during the specific follow-up period after the booster dose.
Occurrence of unsolicited symptoms during the specific follow-up period after the booster dose .
Occurrence of serious adverse events (SAEs) during the entire study period."

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, City of Muntinlupa, Philippines

REFERENCES:
- [Derived] Gatchalian SR, Ramakrishnan G, Bock HL, Lefevre I, Jacquet JM. Immunogenicity, reactogenicity and safety of three-dose primary and booster vaccination with combined diphtheria-tetanus-whole-cell pertussis-hepatitis B-reduced antigen content Haemophilus influenzae type b vaccine in Filipino children. Hum Vaccin. 2010 Aug;6(8):664-72. doi: 10.4161/hv.6.8.12155. PMID 20657177